CLINICAL TRIAL: NCT06485869
Title: Impact of Virtual Reality on the Quality of Life of Oncology Patients
Acronym: VIRONSCARE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Central Hospital Saint Quentin (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2023-A01543-42
Record Dates: First submitted 2024-05-03; First posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-05

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — Quality of Life; Nursing Staff

STUDY DESIGN:
Intervention Model Description: non-randomized parallel two-arm comparative study with a group without virtual reality sessions and a group with virtual reality sessions
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- With virtual reality session (Experimental): Arm A patients will benefit from a 20-minute virtual reality session per chemotherapy session, for the first 3 cycles, with each session lasting more than 30 minutes.
  Interventions: Other: Measure the improvement in quality of life; Other: Measure the level of satisfaction of patients and nursing staff; Other: Measurement of anxiety and pain; Other: Measurement of depressive state; Other: measuring fatigue levels; Other: measurement of acute nausea and vomiting
- Without virtual reality session (Other): Patients in arm B will receive conventional care without hypnotic support.
  Interventions: Other: Measure the improvement in quality of life; Other: Measure the level of satisfaction of patients and nursing staff; Other: Measurement of anxiety and pain; Other: Measurement of depressive state; Other: measuring fatigue levels; Other: measurement of acute nausea and vomiting

INTERVENTIONS:
Other: Measure the improvement in quality of life — Improvment of quality of life is measured by the QLQ-C30 quality of life questionnaire
Other: Measure the level of satisfaction of patients and nursing staff — Patient satisfaction is measured using a five-point scale ranging from 1 = strongly disagree to 5 = strongly agree. Higher scores indicate higher levels of satisfaction.
Other: Measurement of anxiety and pain — Anxiety and pain is measured by Visual Analogue Scale (VAS). This measurement is complemented by physiological responses to anxiety, measured by heart rate and mean arterial blood pressure (HR and BP)
Other: Measurement of depressive state — Depressive State is measured by HAD score
Other: measuring fatigue levels — Fatigue levels is measured by Visual Analogue Scale (VAS).
Other: measurement of acute nausea and vomiting — acute nausea and vomiting is measured by MASCC Antiemesis Tool (MAT)

SUMMARY:
Anxiety, nausea and vomiting are common side effects in paediatric patients receiving chemotherapy. chemotherapy. New evidence supports the efficacy of immersive virtual reality in improving symptoms of anxiety and distress, including nausea and vomiting, in this vulnerable group. This research will evaluate the efficacy of virtual reality in managing anxiety, nausea and vomiting in cancer patients receiving their first line of chemotherapy and will also measure the quality of life of these patients and evaluate patient and nursing staff satisfaction

DETAILED DESCRIPTION:
For cancer patients, virtual reality proved more effective than other forms of distraction in relieving anxiety, depression and fatigue during chemotherapy. Although pain and anxiety in cancer patients are managed proactively, this study was designed to measure the quality of life of these patients, assess patient and carer satisfaction, evaluate the effectiveness of virtual reality in reducing anxiety during the first three sessions of chemotherapy, and assess the impact of virtual reality on preventive and acute chemotherapy-induced fatigue, nausea and vomiting.

This is a clinical study with a therapeutic aim using a non-medicinal, interventional, prospective, multi-centre, controlled and randomised technique, with two parallel groups. It is clinical research involving the human person category 2, involving only minimal risks and constraints. The two arms are Arm A: study questionnaires with virtual reality (VR) Arm B: study questionnaires without virtual reality, standard care (SC)

A visit will be made during the 3 cycles of chemotherapy during which arm A will be immersed in Virtual Reality with the Healthy Mind VR programme.

programme, and patients in arm B will receive standard care without hypnotic support.

There will also be a pre-inclusion visit 7 days before the first cycle. and visits at 3, 6 and 9 months after the 3 cycles of chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Chemotherapy-naive patient
* Patient with first-line indication for intravenous cyclic chemotherapy
* Affiliated to a social security system
* Having received full information on the organization of the research and having given free, informed and written consent signed by the participant and the investigator
* Patient understands French or English
* Expected duration of chemotherapy session for the first 3 cycles greater than 30 minutes

exclusion criteria :

* Patient with communication disorders preventing informed consent
* Patient under legal protection (guardianship, curatorship, safeguard of justice)
* Patients suffering from epilepsy
* Severe visual or hearing impairment preventing use of headphones
* Psychiatric pathologies such as delusional disorders, hallucinations or schizophrenia.
* Patients with infections or facial wounds
* Patients with severe claustrophobia
* Patients with pacemakers
* Patients with known cognitive or learning problems,
* Patients with brain tumors or metastases,
* Patients suffering from motion sickness
* Expected duration of chemotherapy session for the first 3 cycles of 30 minutes or less.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2026-08-29 (Estimated); Study Completion 2026-08-29 (Estimated)

PRIMARY OUTCOMES:
QLQ-C30 | at the start of cycle 1 (each cycle is 28 days); 3,6,9 months post chemo, at the beginning of the 3rd month post chemo, at the beginning of the 6th month post chemo and at the beginning of the 9th month post chemo
  Measurement of the quality of life observed in patients. The QLQ-C30 questionnaire consists of 30 questions on the patient's state of physical and mental health. There are 28 questions with scores ranging from 1 = not at all to 4= very much and two questions with scores ranging from 1= very poor to 7= excellent.
Measuring patient and nurse satisfaction with the chemotherapy procedure | after the first chemotherapy session on day 1 of cycle 1 and 3 (each cycle lasts 28 days)
  Use of a patient questionnaire with a 10-point scale assessed on a five-point scale ranging from 1=strongly disagree disagree to 5 = strongly agree
MAT | after the first chemotherapy session on day 1 of cycle 2 and 3 (each cycle lasts 28 days)
  Assessment of acute nausea and vomiting in patients induced by chemotherapy. 4 questions are used to assess nausea and vomiting 24 hours after chemotherapy and these 4 questions are again used to assess late nausea and vomiting.
  There are 2 questions with a yes or no choice, 1 question with a numerical answer and 1 question with a 10-point numerical scale with 0= none and 10= maximum difficulty.

SECONDARY OUTCOMES:
VAS Score | Before the start of the first chemotherapy session on day 1 of cycle 1, 2 and 3 (each cycle is 28 days) and after the end of the first chemotherapy session on day 1 of cycle 1, 2 and 3 (each cycle is 28 days).
  Measures patients' anxiety and pain levels, as well as their fatigue levels. This questionnaire consists of 4 questions on pain levels, anxiety, fatigue and satisfaction with treatment. It is administered before and after chemotherapy.
  A 10-point numerical scale is used, with 0= the minimum and 10 =the maximum.
Heart rate | Before the start of the first chemotherapy session on day 1 of cycle 1, 2 and 3 (each cycle is 28 days) and after the end of the first chemotherapy session on day 1 of cycle 1, 2 and 3 (each cycle is 28 days).
  Measurement of heart rate in bpm. To assess the patient's level of anxiety and pain. Use of a multiparametric monitor. It will be collected before and after virtual reality.
Blood pressure | Before the start of the first chemotherapy session on day 1 of cycle 1, 2 and 3 (each cycle is 28 days) and after the end of the first chemotherapy session on day 1 of cycle 1, 2 and 3 (each cycle is 28 days).
  Measurement of blood pressure in mmHg. To assess the patient's level of anxiety and pain. Use of a multiparametric monitor. It will be collected before and after virtual reality.
HAD Score | Before the start of the first chemotherapy session on day 1 of cycle 1 (each cycle is 28 days) and after the end of the first chemotherapy session on day 1 of cycle 1 and 2 (each cycle is 28 days).
  Assessment of the patient's state of depression and anxiety. There are 14 questions with scores ranging from 0 to 3 and different answer choices depending on the type of question.

CONTACTS AND LOCATIONS:
Overall Officials: Frédérique Mm Roussel, Principal Investigator — CH SAINT-QUENTIN
Locations (2):
- France (2):
  - Centre Hospitalier de Chauny, Chauny
  - Centre Hospitalier de Saint Quentin, Saint-Quentin

IPD SHARING:
Plan to Share IPD: No
the data will be collected on an electronic Ecrf, a single extraction is planned by the protocol, all the collected data will be analyzed centrally by the study cordernator,no data sharing is planned in the study

REFERENCES:
- [Background] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338
- [Background] Colonna M, Boussari O, Cowppli-Bony A, Delafosse P, Romain G, Grosclaude P, Jooste V; French Network of Cancer Registries (FRANCIM). Time trends and short term projections of cancer prevalence in France. Cancer Epidemiol. 2018 Oct;56:97-105. doi: 10.1016/j.canep.2018.08.001. Epub 2018 Aug 17. PMID 30125884
- [Background] Carnio S, Galetta D, Scotti V, Cortinovis DL, Antonuzzo A, Pisconti S, Rossi A, Martelli O, Cecere FL, Lunghi A, Del Conte A, Montagna ES, Topulli J, Pelizzoni D, Rapetti SG, Gianetta M, Pacchiana MV, Pegoraro V, Cataldo N, Bria E, Novello S. Chemotherapy-induced nausea and vomiting (CINV) in patients with advanced lung cancer during the first-line treatment: assessment by physicians, nurses, and patients from an Italian multicenter survey. Support Care Cancer. 2018 Jun;26(6):1841-1849. doi: 10.1007/s00520-017-4004-1. Epub 2017 Dec 21. PMID 29270827
- [Background] Schneider SM, Workman ML. Effects of virtual reality on symptom distress in children receiving chemotherapy. Cyberpsychol Behav. 1999;2(2):125-34. doi: 10.1089/cpb.1999.2.125. PMID 19178248
- [Background] Chan A, Kim HK, Hsieh RK, Yu S, de Lima Lopes G Jr, Su WC, Banos A, Bhatia S, Burke TA, Keefe DM. Incidence and predictors of anticipatory nausea and vomiting in Asia Pacific clinical practice--a longitudinal analysis. Support Care Cancer. 2015 Jan;23(1):283-91. doi: 10.1007/s00520-014-2375-0. Epub 2014 Aug 13. PMID 25112561
- [Background] Molassiotis A, Lee PH, Burke TA, Dicato M, Gascon P, Roila F, Aapro M. Anticipatory Nausea, Risk Factors, and Its Impact on Chemotherapy-Induced Nausea and Vomiting: Results From the Pan European Emesis Registry Study. J Pain Symptom Manage. 2016 Jun;51(6):987-93. doi: 10.1016/j.jpainsymman.2015.12.317. Epub 2016 Feb 16. PMID 26891606
- [Background] Morrow GR, Roscoe JA, Kirshner JJ, Hynes HE, Rosenbluth RJ. Anticipatory nausea and vomiting in the era of 5-HT3 antiemetics. Support Care Cancer. 1998 May;6(3):244-7. doi: 10.1007/s005200050161. PMID 9629877
- [Background] Dupuis LL, Sung L, Molassiotis A, Orsey AD, Tissing W, van de Wetering M. 2016 updated MASCC/ESMO consensus recommendations: Prevention of acute chemotherapy-induced nausea and vomiting in children. Support Care Cancer. 2017 Jan;25(1):323-331. doi: 10.1007/s00520-016-3384-y. Epub 2016 Aug 26. PMID 27565788
- [Background] Huertas-Fernandez MJ, Martinez-Bautista MJ, Sanchez-Martinez I, Zarzuela-Ramirez M, Baena-Canada JM. [Analysis of the effectiveness of an antiemetic protocol used in an oncology division]. Farm Hosp. 2010 May-Jun;34(3):125-38. doi: 10.1016/j.farma.2009.11.001. Spanish. PMID 20206564
- [Background] Hesketh PJ. Chemotherapy-induced nausea and vomiting. N Engl J Med. 2008 Jun 5;358(23):2482-94. doi: 10.1056/NEJMra0706547. No abstract available. PMID 18525044
- [Background] Birnie KA, Noel M, Parker JA, Chambers CT, Uman LS, Kisely SR, McGrath PJ. Systematic review and meta-analysis of distraction and hypnosis for needle-related pain and distress in children and adolescents. J Pediatr Psychol. 2014 Sep;39(8):783-808. doi: 10.1093/jpepsy/jsu029. Epub 2014 Jun 2. PMID 24891439
- [Background] Vol H, Flank J, Lavoratore SR, Nathan PC, Taylor T, Zelunka E, Maloney AM, Lee Dupuis L. Poor chemotherapy-induced nausea and vomiting control in children receiving intermediate or high dose methotrexate. Support Care Cancer. 2016 Mar;24(3):1365-71. doi: 10.1007/s00520-015-2924-1. Epub 2015 Sep 3. PMID 26335406
- [Background] Ovayolu N, Ovayolu O, Serce S, Tuna D, Pirbudak Cocelli L, Sevinc A. Pain and quality of life in Turkish cancer patients. Nurs Health Sci. 2013 Dec;15(4):437-43. doi: 10.1111/nhs.12047. Epub 2013 Mar 11. PMID 23480371
- [Background] Ahmed RL, Prizment A, Lazovich D, Schmitz KH, Folsom AR. Lymphedema and quality of life in breast cancer survivors: the Iowa Women's Health Study. J Clin Oncol. 2008 Dec 10;26(35):5689-96. doi: 10.1200/JCO.2008.16.4731. Epub 2008 Nov 10. PMID 19001331
- [Background] Dupuis LL, Robinson PD, Boodhan S, Holdsworth M, Portwine C, Gibson P, Phillips R, Maan C, Stefin N, Sung L; Pediatric Oncology Group of Ontario. Guideline for the prevention and treatment of anticipatory nausea and vomiting due to chemotherapy in pediatric cancer patients. Pediatr Blood Cancer. 2014 Aug;61(8):1506-12. doi: 10.1002/pbc.25063. Epub 2014 Apr 17. PMID 24753095
- [Background] Chirico A, Lucidi F, De Laurentiis M, Milanese C, Napoli A, Giordano A. Virtual Reality in Health System: Beyond Entertainment. A Mini-Review on the Efficacy of VR During Cancer Treatment. J Cell Physiol. 2016 Feb;231(2):275-87. doi: 10.1002/jcp.25117. PMID 26238976
- [Background] Wong CL, Ip WY, Kwok BMC, Choi KC, Ng BKW, Chan CWH. Effects of therapeutic play on children undergoing cast-removal procedures: a randomised controlled trial. BMJ Open. 2018 Jul 5;8(7):e021071. doi: 10.1136/bmjopen-2017-021071. PMID 29980545
- [Background] Chan CW, Lam LW, Li CK, Cheung JS, Cheng KK, Chik KW, Chan HY, So WK, Tang WP. Feasibility of psychoeducational interventions in managing chemotherapy-associated nausea and vomiting (CANV) in pediatric oncology patients. Eur J Oncol Nurs. 2015 Apr;19(2):182-90. doi: 10.1016/j.ejon.2014.09.002. Epub 2014 Oct 25. PMID 25445732
- [Background] Rutter CE, Dahlquist LM, Weiss KE. Sustained efficacy of virtual reality distraction. J Pain. 2009 Apr;10(4):391-7. doi: 10.1016/j.jpain.2008.09.016. Epub 2009 Feb 23. PMID 19231295
- [Background] Schneider SM, Kisby CK, Flint EP. Effect of virtual reality on time perception in patients receiving chemotherapy. Support Care Cancer. 2011 Apr;19(4):555-64. doi: 10.1007/s00520-010-0852-7. Epub 2010 Mar 26. PMID 20336327
- [Background] Schneider SM, Hood LE. Virtual reality: a distraction intervention for chemotherapy. Oncol Nurs Forum. 2007 Jan;34(1):39-46. doi: 10.1188/07.ONF.39-46. PMID 17562631
- [Background] Schneider SM, Workman ML. Virtual reality as a distraction intervention for older children receiving chemotherapy. Pediatr Nurs. 2000 Nov-Dec;26(6):593-7. PMID 12026359
- [Background] Karaman D, Erol F, Yilmaz D, Dikmen Y. Investigation of the effect of the virtual reality application on experimental pain severity in healthy. Rev Assoc Med Bras (1992). 2019 Mar;65(3):446-451. doi: 10.1590/1806-9282.65.3.446. Epub 2019 Apr 11. PMID 30994846
- [Background] Zeng Y, Zhang JE, Cheng ASK, Cheng H, Wefel JS. Meta-Analysis of the Efficacy of Virtual Reality-Based Interventions in Cancer-Related Symptom Management. Integr Cancer Ther. 2019 Jan-Dec;18:1534735419871108. doi: 10.1177/1534735419871108. PMID 31441352
- [Background] Bani Mohammad E, Ahmad M. Virtual reality as a distraction technique for pain and anxiety among patients with breast cancer: A randomized control trial. Palliat Support Care. 2019 Feb;17(1):29-34. doi: 10.1017/S1478951518000639. Epub 2018 Sep 10. PMID 30198451
- [Background] Chirico A, Maiorano P, Indovina P, Milanese C, Giordano GG, Alivernini F, Iodice G, Gallo L, De Pietro G, Lucidi F, Botti G, De Laurentiis M, Giordano A. Virtual reality and music therapy as distraction interventions to alleviate anxiety and improve mood states in breast cancer patients during chemotherapy. J Cell Physiol. 2020 Jun;235(6):5353-5362. doi: 10.1002/jcp.29422. Epub 2020 Jan 20. PMID 31957873
- See also: The prevalence of long-term symptoms of depression and anxiety after breast cancer treatment: A systematic review — https://doi.org/10.1016/j.maturitas.2015.04.010
- See also: Projection de l'incidence et de la mortalité par cancer en France métropolitaine en 2017 — https://www.santepubliquefrance.fr/docs/projection-de-l-incidence-et-de-la-mortalite-par-cancer-en-france-metropolitaine-en-2017